CLINICAL TRIAL: NCT02898376
Title: Evaluation of the Clinical Benefit of a Spa Care on the Evolution of Late Fibrosis After Postoperative Radiotherapy for Breast Cancer in Remission
Brief Title: Clinical Benefit of Spa Care on Severe Radiation-induced Fibrosis After Postoperative Radiotherapy for Breast Cancer
Acronym: FIBROTHERME
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut de Cancérologie de Lorraine (Other)
Collaborators: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-003518-28
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Breast Carcinoma; Fibrosis
Keywords: spa care; randomised controlled trial; pentoxifylline/tocopherol combination; late sequelae; radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Fibrosis | interventions — Pentoxifylline; alpha-Tocopherol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination tocopherol/pentoxifylline + spa care (Experimental): pentoxifylline (400 mg bid) + tocopherol (500 mg x bid) during at least 6 months AND skin-oriented spa care (18 days)
  Interventions: Other: skin-oriented spa care; Drug: Pentoxifylline; Drug: Tocopherol acetate
- combination tocopherol/pentoxifylline (Active Comparator): pentoxifylline (400 mg bid) + tocopherol (500 mg x bid) during at least 6 months
  Interventions: Drug: Pentoxifylline; Drug: Tocopherol acetate

INTERVENTIONS:
Other: skin-oriented spa care — standardized procedure : 72 care sessions over 18 days of treatment
  +/- Additional care according to the specificity of each spa
  Arms: combination tocopherol/pentoxifylline + spa care
Drug: Pentoxifylline — 400 mg bid during at least 6 months
Drug: Tocopherol acetate — 500 mg bid during at least 6 months

SUMMARY:
This study evaluates the dermatological life quality six months after spa cares in patients with severe late toxicity involving the skin and / or soft tissues after postoperative radiotherapy for breast cancer. Half of the patients will be treated with a combination of pentoxifylline (PTX) and alpha-tocopherol (Vit E) when Half of the patients will receive skin-oriented spa cares in addition.

DETAILED DESCRIPTION:
The combination of PTX and vit E appears as the standard treatment of radiation induced fibrosis. Synergism between PTX and Vit E is likely, as treatment with each drug alone is ineffective. This combination was also positively evaluated in the treatment of osteoradionecrosis, radiation-induced pelvic neuropathies, pneumoniae as well as bowel pathologies.

Spa cares are part of the standard treatment of burn scars. Two spa treatments per year enable the mitigation or disappearance (after several treatments) of pruritus, dysesthesia, local inflammation, hypertrophy and sclerosis. They promote the healing of chronic superficial erosions. The spa treatment combines baths, sprays and especially filiform showers with thermal water jets under high pressure for a few minutes.

ELIGIBILITY:
Inclusion Criteria:

* women
* age ≥ 18 and <80 years old
* invasive or in situ breast carcinoma
* non-metastatic disease.
* postoperative radiotherapy completed since at least 6 months
* unilateral breast radiotherapy
* grade > 2 dermal and/or soft tissue toxicity (CTCAE v4.0)
* no inflammatory ou infectious flare on the breast at the time of inclusion
* ability to provide an informed written consent form
* affiliation to a social security system

Exclusion Criteria:

* age <18 or ≥ 80 years old
* evolutive cancer
* Metastatic Disease
* Patient undergoing specific treatment for breast cancer (except adjuvant endocrine therapy and / or adjuvant Herceptin) at the time of inclusion
* bilateral Breast/chest wall Radiotherapy
* breast prosthesis bearer
* Body Mass Index > 40 or <18.5
* chronic skin ulceration within the treated breast at the time of inclusion
* contraindications to spa care :

  * inflammatory disease in flare at the time of inclusion
  * active infections
  * heart failure (NYHA class> 1)
  * chronic respiratory failure
  * labile blood pressure
  * bullous dermatitis
* evolutive chronic skin disease
* hypersensitivity to pentoxifylline or any of the excipients
* acute myocardial infarction
* ongoing hemorrhage or major bleeding risk
* use of oral anticoagulants
* pregnant or likely to be in 6 months or breastfeeding
* patients deprived of liberty or under supervision

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Dermatology Quality of life at 6 months | 6 months after the end of treatment
  Self-reported dermatology quality of life using the standardized Dermatology Life Quality Index (DLQI) ; This score assess the functional impact of fibrosis: eg. intensity of pain, itching... (10 items). The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.

SECONDARY OUTCOMES:
Dermatology Quality of life at 12 months | 12 months after the end of treatment
  Self-reported dermatology quality of life using the standardized Dermatology Life Quality Index (DLQI) ; This score assess the functional impact of fibrosis: eg. intensity of pain, itching... (10 items). The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Overall quality of life | 6 months
  quality of life questionnaire (EORTC QLQ C30 score)
Breast-oriented quality of life | 6 months
  EORTC QLQ-BR23 score
late radiation toxicity | 6 months
  Evaluation of late toxicity performed independently and in blind by another radiation oncologist from the same center, using the CTCAE v4.0 scale modules: Skin and subcutaneous tissue disorders / Musculoskeletal skeletal / Reproductive organs and breast
Skin thickness | 6 months
  The skin thickness will be assessed in blind by an independently radiologist using a standardized Ultrasound scan procedure (Yoshida EJ, et al; Int J Radiat Oncol Biol Phys. 2012) Skin thickness is measured as the distance between the entry ultrasound echo signal to the border between the dermis and hypodermis . Measurements are acquired from ten locations: five on the treated (irradiated) breast (12:00, 3:00, 6:00, 9:00, and tumor bed), and five corresponding locations on the untreated (contralateral) breast - serving as controls to account for patient baseline variation
Cosmetic appearance | 6 months
  The cosmetic appearance will be evaluated by the investigator with the Harvard-breast-cosmesis-scale (HBCS). HBCS classifies the overall aesthetic results in four categories from excellent, good, fair to poor; comparing the treated breast to the control breast

CONTACTS AND LOCATIONS:
Overall Officials: VOGIN Guillaume, MD,PhD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (21):
- France (21):
  - CHU de Besançon Hôpital Jean Minjoz, Besançon
  - ONCODOC, Béziers
  - Centre d'Oncologie et de Radiothérapie du Parc, Chalon-sur-Saône
  - Clinique du Parc de Charleville-Mézières, Charleville-Mézières
  - CLCC Jean Perrin, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - Centre Georges-François Leclerc, Dijon
  - Institut Daniel Hollard, Grenoble
  - CHU de Grenoble, Hôpital A.Michallon, La Tronche
  - CHR Metz-Thionville Hôpital de Mercy, Metz
  - CH de Belfort-Montbéliard Site du Mittan, Montbéliard
  - CH de Mulhouse, Mulhouse
  - Centre d'Oncologie de Gentilly, Nancy
  - CHU de Poitiers, Poitiers
  - Institut Jean Godinot de Reims, Reims
  - CLCC Saint Etienne, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Clinique de l'Orangerie, Strasbourg
  - Institut Universitaire du Cancer, Toulouse
  - CH de Troyes, Troyes
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No